CLINICAL TRIAL: NCT00166400
Title: Beta Blockade in Mitral Regurgitation
Brief Title: A Randomized Clinical Trial of Metoprolol in Participants With Mitral Regurgitation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Maurice Sarano, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 960-04; IRUSMETO0047, IRB 960-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: metoprolol succinate — Treatment with potent beta-blockade titrated to the maximally tolerated dose.

SUMMARY:
Mitral valve regurgitation (leakage of the mitral valve of the heart) is frequent and currently there is no specific medical therapy. Mitral regurgitation is a slowly progressive disease that frequently requires surgical treatment. This randomized clinical trial will use Metoprolol, a common beta-blocker medication, to determine if medical treatment impacts mitral valve disease progression.

DETAILED DESCRIPTION:
Background: Mitral regurgitation (MR) is frequent and its prevalence is increasing with aging of the population. Organic MR, due to primary valvular lesions has severe consequences determined by its degree, with left ventricular (LV) remodeling and dysfunction, left atrial (LA) enlargement, leading to poor clinical outcome. Surgery can eliminate MR, but carries notable risks and is not applicable to all patients. Recent animal data suggest that beta-blockade in organic MR has significant positive effect, particularly on LV remodeling. Therefore, chronically decreasing MR, protecting LV and LA with beta-blockade are major goals of medical therapy. However, effects of chronic oral beta-blockade of human MR are uncertain and recent practice guidelines underscored these gaps in knowledge and did not recommend beta-blockade of MR. Hence, a trial of treatment of organic MR is needed. A large trial with mortality-morbidity end-points is desirable but premature without knowledge of magnitude of mechanistic effects of beta-blockade. The improvement of these intermediate end-points, mechanistically linked to outcome, is measurable with non-invasive quantitative techniques and forms the basis of the present clinical trial proposal. Hypothesis: Chronic beta-blockade therapy using Metoprolol weighed against placebo produces a sustained reduction of the consequences of organic MR. Specific aims are that treatment improves a) degree of MR (decreases regurgitant volume, primary end-point), b) LV remodeling (decreases LV end-diastolic volume index, second end-point), and c) LA enlargement (decreases LA volume, third end-point) as compared to placebo. Population: Patients with MR organic (intrinsic valve disease), isolated (no other valve disease) d moderate (regurgitant volume *30 mL/beat). Methods: A randomized clinical trial, placebo controlled, double-blind, without crossover, of 12 months oral treatment with potent beta-blockade (Metoprolol XL 50 to 200mg QD) titrated to the maximally tolerated dose. The trial is preceded by an acute study to determine tolerance. End-points are measured by Doppler-Echocardiography for quantitation of MR (regurgitant volume) using combination of 3 simultaneous methods (quantitative Doppler, two-dimensional echocardiography, proximal flow convergence) and echocardiography for LV and LA volume measurement. In addition cardiopulmonary exercise testing will measure peak O2 consumption at baseline and follow-up. This study seeks to enroll a total of 60 patients. The analysis will be based on intention to treat and compare changes in regurgitant volume, LV end-diastolic volume index and LA volume measured after one year of treatment with active drug or placebo. The results of this clinical trial should provide strong evidence regarding medical treatment of patients with organic MR and define future strategies to minimize mortality and morbidity of organic MR.

ELIGIBILITY:
Inclusion criteria: Patients a) 21 years old or older, with b) MR observed with color flow imaging, c) due to organic mitral valve disease demonstrated by Echocardiography (not normal valve as in functional or ischemic MR), c) isolated (no valve disease other than functional tricuspid regurgitation by Doppler-Echocardiography), d) pure (no mitral stenosis by Doppler-Echocardiography), e) quantifiable by Doppler-Echocardiography, f) of degree * moderate, defined as RVol * 30 mL/beat, g) occurring on native valves, h) with echocardiographic imaging allowing assessment of LA and LV, and i) asymptomatic (or mildly symptomatic but not considered as candidates for immediate surgery by their attending physician).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Degree of mitral regurgitation, assessed as the regurgitant volume, at baseline and 12 months | baseline & 12 months

SECONDARY OUTCOMES:
Left ventricular end-diastolic volume index at baseline and 12 months | baseline & 12 months
Left atrial end-diastolic volume at baseline and at 12 months | baseline & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurice E Sarano, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States